CLINICAL TRIAL: NCT07056725
Title: Quality of Life and Sleep in Patients With Temporomandibular Disorders. A Protocol for a Randomized Control Trial
Brief Title: Quality of Life and Sleep in Patients With Temporomandibular Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Clinical Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIM/2025/3
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Temporomandibular Disorders (TMDs)
Keywords: Manual Therapy; Therapeutic Exercise; Quality of life; Quality of Sleep
MeSH Terms: conditions — Temporomandibular Joint Disorders; Sleep Initiation and Maintenance Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: An experimental study is proposed in the form of a Randomized Controlled Trial (RCT), longitudinal and prospective in design, with two intervention groups.
  Patients with Temporomandibular Disorders (TMD) will be randomly assigned to two intervention groups (G1 and G2), ensuring that participants in both groups present with similar baseline characteristics.
  The 25 requirements proposed by the CONSORT declaration will be followed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Subjects in this group will receive physiotherapy treatment consisting of a Manual Therapy program targeting the orofacial region, combined with a Cervical Therapeutic Exercise program. The Cervical Therapeutic Exercise program focuses on co-contraction exercises of the flexor and extensor muscles, progressively increasing difficulty and resistance through the use of a latex band (Theraband), along with neural tissue techniques.
  Interventions: Other: Manual Therapy and Therapeutic Exercises Programs
- Group 2 (Experimental): Subjects in this group will receive physiotherapy treatment consisting of a Manual Therapy program targeting the orofacial region, combined with an Orofacial Therapeutic Exercise program. The Orofacial Therapeutic Exercise program focuses on coordination exercises of the masseter muscles, progressively increasing difficulty and resistance, and is combined with neural tissue techniques.
  Interventions: Other: Manual Therapy and Therapeutic Exercises Programs

INTERVENTIONS:
Other: Manual Therapy and Therapeutic Exercises Programs — A treatment based on the combination of Manual Therapy targeting the orofacial region and a therapeutic exercise program focused on either the cervical or orofacial region

SUMMARY:
The aim of this study is to evaluate and compare the effects of two physiotherapeutic intervention programs on the quality of life in patients with Temporomandibular Disorders (TMD).

Study design: Randomized, longitudinal, and prospective clinical trial with two intervention groups.

Population: Subjects aged 18-65 years with subacute temporomandibular disorders.

DETAILED DESCRIPTION:
The study will be carried out at the Faculty of Nursing and Physiotherapy of the University of Alcalá. A total of 30 subjects with Temporomandibular Disorders (TMD) will be selected and randomly assigned into two intervention groups.

The first group will receive a physiotherapy treatment based on a Manual Therapy program targeting the orofacial region, combined with a Cervical Therapeutic Exercise program. In contrast, the second group will receive a physiotherapy treatment based on a Manual Therapy program for the orofacial region, combined with an Orofacial Therapeutic Exercise program.

Both groups will undergo a total of six treatment sessions over a period of six weeks (1 session per week). Each manual therapy session targeting the orofacial region will last 30 minutes. The manual therapy (MT) techniques will include a combination of neuromuscular and articular manual techniques.

The study will assess the following variables: quality of life, sleep quality, pressure pain threshold, maximum pain-free mouth opening, perceived pain, and treatment adherence.

Measurements will be taken pre-treatment, post-treatment and a follow-up at 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years of age with subacute Temporomandibular Disorders (TMD).
* Diagnosis of TMD based on: The Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). And The Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD).
* Willingness to participate in the study and signing of the informed consent form.

Exclusion Criteria:

* Individuals younger than 18 years or older than 65 years.
* Medical history or systemic conditions, including: Diagnosis of neurological or neuromuscular disorders (such as multiple sclerosis, facial paralysis, trigeminal neuralgia). Systemic or inflammatory joint diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, fibromyalgia). Presence of severe psychiatric disorders. Previous diagnosis of cancer in the craniofacial or cervical region.
* Previous interventions (e.g., surgery involving the TMJ or the orofacial and cervical regions).
* History of trauma in the region, including mandibular trauma, whiplash injuries, or fractures in the area.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (SF-12) | Pre-intervention, post-intervention (6 weeks) and follow-up of 8 weeks after the end
  The SF-12 consists of a subset of 12 items from the SF-36, covering physical functioning, social functioning, physical role, emotional role, mental health, vitality, bodily pain, and general health. The SF-12 is a shortened version of the SF-36 Health Survey. It is a self-administered questionnaire with a completion time of less than 2 minutes. The response options are based on Likert-type scales that assess intensity or frequency. The number of response options ranges from three to six, depending on the item.
Sleep Quality (Pittsburgh Sleep Quality Index) | Pre- intervation, post-intervention (6 weeks) and follow-up of 8 weeks after the end.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-administered instrument designed to assess sleep quality in adults over the past month. It consists of 19 items grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.

SECONDARY OUTCOMES:
Pain Intensity (NRS) | Pre- intervention, post- intervention (6 weeks) and follow-up of 8 weeks after the end
  The Numerical Rating Scale (NRS) is a widely used instrument for the subjective assessment of pain intensity.
  It consists of a numerical scale from 0 to 10, where 0 indicates no pain and 10 represents the highest intensity. Patients select the number that best reflects the severity of their symptom.
Pressure Pain Threshold (PPT) | Pre- intervention, post- interventio (6 weeks) and follow-up of 8 weeks after the end.
  The tip of the algometer will be applied perpendicularly to the muscle (anterior portion of the temporalis muscle and the superficial belly of the masseter muscle), and pressure will be gradually increased at a rate of 1 kg/sec. Participants will be instructed to signal the moment they first perceive pain, in order to accurately record the pressure pain threshold.
Maximum Pain-Free Mouth Opening (MPMO) | Pre- intervention, post- intervention (6 weeks) and follow-up of 8 weeks after the end.
  MPMO is a clinical measure used to assess mandibular function in patients with temporomandibular disorders (TMD). This variable evaluates the ability to open the mouth without experiencing pain, reflecting the functional status of the temporomandibular joint and the associated musculoskeletal structures.
Treatment Adherence | Post- intervention (6 weeks)
  A personalized diary will be provided for each participant in both groups. Each program will include an exercise log that patients will be required to complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Alcalá De Henares, Madrid, Alcalá de Henares, Spain

IPD SHARING:
Plan to Share IPD: No